CLINICAL TRIAL: NCT03046849
Title: Diagnosis of Lynch Syndrome Based on Next-generation Sequencing in Colorectal Cancer Patients Meeting Chinese Lynch Syndrome Criteria: An Open-label and Multi-center Study.
Brief Title: Diagnosis of Lynch Syndrome Based on Next-generation Sequencing in Patients Meeting Chinese Lynch Syndrome Criteria
Status: Completed | Type: Observational
Sponsor: Second Affiliated Hospital, School of Medicine, Zhejiang University (Other)
Responsible Party: Principal Investigator, Ying Yuan, MD, Professor, Department of Medical Oncology, Second Affiliated Hospital, School of Medicine, Zhejiang University
Other Study IDs: HDLS201701
Record Dates: First submitted 2017-02-06; First posted 2017-02-08 (Estimated); Last update posted 2021-08-11 (Actual); Status verified 2017-02

CONDITIONS: Lynch Syndrome
Keywords: Lynch Syndrome; next-generation sequencing; germline mutation
MeSH Terms: conditions — Colorectal Neoplasms, Hereditary Nonpolyposis | interventions — High-Throughput Nucleotide Sequencing

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — whole blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: next-generation sequencing — Use next-generation sequencing to test germline mutation.

SUMMARY:
The purpose of this study is to find out the proportion of patients diagnosed with Lynch syndrome in colorectal cacner patients meeting Chinese Lynch syndrome criteria. Besides, this study is aimed to analyze the clinical characteristics and germline mutation of Lynch syndrome in Chinese population.

DETAILED DESCRIPTION:
1. Detect germline mutation (by next-generation squencing) in probands.
2. Verify the germline mutation in blood relatives whose proband has known germline mutation(s).
3. Analyze the test data with clinical and family information. Diagnose Lynch syndrome in the included population.
4. Analyze the clinical characteristics and germline mutation of Lynch syndrome in Chinese population.

ELIGIBILITY:
For probands, the inclusion criteria： all of the following three points should be satisfied:

1. One of the colorectal cancer patients from families meeting Chinese Lynch syndrome criteria.

   Chinese Lynch syndrome criteria:

   In a pedigree, there were at least 2 patients with histological-proven colorectal cancer, and among these, at least two patients are first-degree relatives of each other. Besides, any one of the following three points should be satisfied in the pedigree:

   A. at least one patients with multiple primary colorectal carcinoma/adenoma, either synchronously or metachronously.

   B. at least one colorectal cancer diagnosed before 50 years old. C. in the pedigree, at least one patient diagnosed with other Lynch syndrome associated cancer (ie, gastric, endometrial, small bowel, ureter, or renal-pelvic, ovarian and hepatobiliary cancers).
2. With sufficient blood to test;
3. Agree to provide basic information, clinical information and family history of cancer information.

For probands, the exclusion criteria:

With at least one blood relative with known pathogenic germline mutation(s).

For blood relatives verifying germline mutation, the inclusion criteria： all of the following three points should be satisfied:

1. First- to second-degree blood relatives of probands with germline mutation(s).
2. With sufficient blood to test.
3. Agree to provide basic information, clinical information and family history of cancer information.

For blood relatives verifying germline mutation, the exclusion criteria:

Blood relatives who refuse to test.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: The probands will be selected from colorectal cancer patients meeting Chinese Lynch syndrome criteria. The blood relatives verifying germline mutation will be selected from whose proband has germline mutation(s).
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2017-03-08 (Actual); Primary Completion 2019-02-26 (Actual); Study Completion 2019-02-26 (Actual)

PRIMARY OUTCOMES:
Pathogenic germline mutation | Upon completion of study, on average 2 years.
  Pathogenic germline mutation using next-generation sequencing with a targeted panel.

SECONDARY OUTCOMES:
Variant of uncertain significance of germline mutation | Upon completion of study, on average 2 years.
  Variant of uncertain significance using next-generation sequencing with a targeted panel.

CONTACTS AND LOCATIONS:
Overall Officials: Ying Yuan, Ph.D, MD, Principal Investigator — Second Affiliated Hospital, School of Medicine, Zhejiang University
Locations (3):
- China (3):
  - Jiangsu Province Hospital, Nanjing, Jiangsu
  - West China Hospital, Chengdu, Sichuan
  - The second affiliated hospital of Zhejiang University, Hangzhou, Zhejinag

IPD SHARING:
Plan to Share IPD: Undecided